CLINICAL TRIAL: NCT03013114
Title: A Single-center Clinical Trial of Bortezomib in Management of Immune Thrombocytopenia (ITP) With High Anti-platelet Antibodies Level
Brief Title: A Single-center Clinical Trial of Bortezomib in Management of Immune Thrombocytopenia (ITP)
Acronym: ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Bortezomib
Record Dates: First submitted 2016-12-22; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Immune Thrombocytopenia
Keywords: Bortezomib Immune thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Experimental): Bortezomib was given by intravenous bolus injection at a dose of 1.3 mg/m2 on days 1, 4, 8 and 11, repeated every 21 days. It will be given four cycles.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib was given by intravenous bolus injection at a dose of 1.3 mg/m2 on days 1, 4, 8 and 11, repeated every 21 days. It will be given four cycles.

SUMMARY:
Primary immune thrombocytopenia (ITP) is a disorder caused by autoantibody-mediated platelet destruction and decreased platelet production. It has been reported that refractory ITP is closely related to long-lived plasma cells (PCs), which are resistant to glucocorticoids, conventional immunosuppressive and cytotoxic drugs, irradiation and B-cell depletion therapies.

Proteasome inhibition bortezomib is one of the most promising therapeutic approaches to target PCs, since this strategy has been shown to efficiently eliminate multiple myeloma cells, that is, transformed PCs. It also has been successfully used in SLE-like mice, experimental autoimmune MG rats and experimental hemophilia-A mice that develop anti-factor VIII antibodies in preclinical models by depleting both short-lived and long-lived PCs. Additionally, treatment with bortezomib resulted in a rapid clinical response in a patient with refractory thrombotic thrombocytopenic purpura associated with the depletion of inhibitory autoantibodies against ADAMTS13, a metalloproteinase that cleaves the von Wille-brand factor, which is produced by plasma cells. Hence, the elimination of autoreactive PCs by proteasome inhibitors might represent a new treatment strategy for autoantibody-mediated diseases.

To date, refractory ITP is lacking of effective treatments and these findings encouraged us to conduct a study of bortezomib in management of ITP with high anti-platelet antibodies level. Data from this study may provide some idea of bortezomib in the treatment of ITP.

DETAILED DESCRIPTION:
The investigators are undertaking a single-center, single-arm study of 20 primary ITP adult patients from Shandong University Qilu Hospital

. All the participants are selected to receive bortezomib treatment (given intravenously at a dose of 1.3mg/m2 on days 1,4,8,11). Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* failure to achieve at least Response
* need of treatment(s) (including, but not limited to, low dose of corticosteroids) to minimize the risk of clinically significant bleeding. Need of on-demand or adjunctive therapy alone does not qualify the patient as refractory
* primary ITP confirmed by excluding other supervened causes of thrombocytopenia

Exclusion Criteria:

* pregnancy
* hypertension
* cardiovascular disease
* diabetes
* liver and kidney function impairment
* HCV, HIV, HBsAg seropositive status
* patients with systemic lupus erythematosus and/or antiphospholipid syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Platelet counts | an average of 3 months
  1. Complete response (CR)： A platelet count ≥ 100 * 10^9/L measured on two occasions > 7 days apart and the absence of bleeding.
  2. Response (R)： A platelet count ≥ 30 * 10^9/L and a greater than two fold increase in platelet count from baseline measured on two occasions > 7 days apart and the absence of bleeding.
  3. No response (NR)： A platelet count < 30 * 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

SECONDARY OUTCOMES:
Numbers of Megakaryocyte Polyploidy | 6 days after every treatment cycle, an average of 3 months
Expression rate of long-lived plasma cells | 6 days after every treatment cycle, an average of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Shandong University Qilu hospital, Jinan, Shandong, China